CLINICAL TRIAL: NCT02737501
Title: A Phase 3 Multicenter Open-label Study of Brigatinib (AP26113) Versus Crizotinib in Patients With ALK-positive Advanced Lung Cancer
Brief Title: ALTA-1L Study: A Study of Brigatinib Versus Crizotinib in Anaplastic Lymphoma Kinase Positive (ALK+) Advanced Non-small Cell Lung Cancer (NSCLC) Participants
Acronym: ALTA-1L
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP26113-13-301; U1111-1210-4363 (Other: WHO); 2015-003447-19 (EudraCT Number)
Record Dates: First submitted 2016-03-30; First posted 2016-04-14 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer; Advanced Malignancies; Carcinoma
Keywords: Non-small cell lung cancer; Non-small cell lung carcinoma; Epithelial lung cancer; Squamous cell carcinoma; Large cell carcinoma; Adenocarcinoma; Carcinoma; Anaplastic Lymphoma Kinase (ALK); Advanced Cancers; Brigatinib; AP26113
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma; Carcinoma, Squamous Cell; Carcinoma, Large Cell; Adenocarcinoma | interventions — brigatinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Randomized Phase: Brigatinib 90 mg QD/180 QD (Experimental): Brigatinib 90 mg, tablets, orally, QD for first 7 days followed by 180 mg, orally, QD, in each 28-day cycle until PD, intolerable toxicity, consent withdrawal, or death (The median duration of exposure was 34.86 months).
  Interventions: Drug: Brigatinib
- Randomized Phase: Crizotinib 250 mg BID (Active Comparator): Crizotinib 250 mg, tablets, BID in each 28-day cycle until disease progression, intolerable toxicity, consent withdrawal, or death (The median duration of exposure was 9.26 months).
  Interventions: Drug: Crizotinib
- Crossover Phase: Brigatinib 90 mg QD/180 mg QD (Experimental): Participants who experienced PD as assessed by the BIRC or received radiotherapy to the brain while on 'Crizotinib 250 mg BID' therapy in Randomized Phase were crossed over. Following 10-day washout period, crossover participants received brigatinib 90 mg, tablets, orally, QD for first 7 days followed by 180 mg, tablets, orally, QD in each 28-day cycle up to end of the study (The median duration of exposure was 17.25 months).
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib tablets
  Arms: Crossover Phase: Brigatinib 90 mg QD/180 mg QD; Randomized Phase: Brigatinib 90 mg QD/180 QD
Drug: Crizotinib — Crizotinib tablets
  Other Names: Xalkori
  Arms: Randomized Phase: Crizotinib 250 mg BID

SUMMARY:
The purpose of the study is to compare the efficacy of brigatinib to that of crizotinib in ALK+ locally advanced or metastatic non-small cell lung cancer (NSCLC) participants naive to ALK inhibitors, as evidenced by progression-free survival (PFS).

DETAILED DESCRIPTION:
The purpose of this phase III, randomized, open-label, comparative, multicenter, international study is to compare the efficacy and safety of brigatinib to that of crizotinib in ALK+ locally advanced or metastatic NSCLC participants who have not previously been treated with an ALK inhibitor. Participants will be stratified by the presence of CNS metastases at baseline and prior chemotherapy used for locally advanced or metastatic disease. Participants will be randomized in a 1:1 ratio to receive either brigatinib, 90 mg orally once daily (QD) for 7 days, then a 180 mg orally QD, or crizotinib, 250 mg orally twice daily (BID). Participants will receive treatment until disease progression, intolerable toxicity, consent withdrawal, or death. Crossover from crizotinib to brigatinib is also permitted.

The total estimated duration of the study is at least 4.5 years, including 1.5 years to accrue participants, with at least 3 years for treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed stage IIIB (and not a candidate for definitive multimodality therapy) or stage four (IV) NSCLC.
2. Must have documented ALK rearrangement.
3. Have sufficient tumor tissue available for central analysis.
4. Have at least 1 measurable (that is, target) lesion per RECIST v1.1.
5. Recovered from toxicities related to prior anticancer therapy to National Cancer Institute (of the United States) (NCI) Common Terminology Criteria for Adverse Events (version 4.0) (CTCAE v 4.0) grade be less than or equal to (<=) 1.
6. Are a male or female participants greater than or equal to (>=)18 years old.
7. Have adequate organ function, as defined by the study protocol.
8. Have Eastern Cooperative Oncology Group (ECOG) performance status <=2.
9. Have normal QT interval on screening ECG evaluation, defined as QT interval corrected (Fridericia) (QTcF) of <= 450 millisecond (msec) in males or <=470 msec in females.
10. For female participants of childbearing potential, have a negative pregnancy test documented prior to randomization.
11. For female and male participants who are fertile, agree to use a highly effective form of contraception, as defined by the study protocol.
12. Provide signed and dated informed consent indicating that the participants has been informed of all pertinent aspects of the study, including the potential risks, and is willingly participating.
13. Have the willingness and ability to comply with scheduled visit and study procedures.

Exclusion Criteria:

1. Previously received an investigational antineoplastic agent for NSCLC.
2. Previously received any prior tyrosine kinase inhibitor (TKI), including ALK-targeted TKIs.
3. Previously received more than 1 regimen of systemic anticancer therapy for locally advanced or metastatic disease.
4. Received chemotherapy or radiation within 14 days of first dose of study drug, except stereotactic radiosurgery (SRS) or stereotactic body radiation therapy (SBRT).
5. Received anti-neoplastic monoclonal antibodies within 30 days of the first dose of study drug.
6. Had major surgery within 30 days of the first dose of study drug, minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.
7. Have been diagnosed with another primary malignancy other than NSCLC, except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or participants with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
8. Have symptomatic CNS metastases (parenchymal or leptomeningeal) at screening or asymptomatic disease requiring an increasing dose of corticosteroids to control symptoms within 7 days prior to randomization.
9. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Participants with leptomeningeal disease and without cord compression are allowed.
10. Be pregnant, planning a pregnancy, or breastfeeding.
11. Have significant, uncontrolled, or active cardiovascular disease, as defined by the study protocol.
12. Have uncontrolled hypertension.
13. Have a history or the presence at baseline of pulmonary interstitial disease, drug-related pneumonitis, or radiation pneumonitis.
14. Have an ongoing or active infection.
15. Have a known history of human immunodeficiency virus (HIV) infection.
16. Have a known or suspected hypersensitivity to brigatinib or its excipients and/or crizotinib or its excipients.
17. Have malabsorption syndrome or other gastrointestinal (GI) illness or condition.
18. Have any condition or illness that, in the opinion of the investigator, would compromise participant's safety or interfere with the evaluation of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (91):
- United States (12):
  - USOR - Arizona Oncology Associates - Sedona, Sedona, Arizona
  - Kaiser Permanente Bellflower Medical Offices, Bellflower, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Boulder, Boulder, Colorado
  - Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Minnesota Oncology, Coon Rapids, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Oncology Hematology Care - Blue Ash, Cincinnati, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
- Australia (4):
  - Saint George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Monash Medical Centre, Bentleigh East, Victoria
  - Saint Vincent's Hospital Melbourne, Fitzroy, Victoria
- Austria (2):
  - Universitatsklinium St. Polten, Sankt Pölten, Lower Austria
  - Otto-Wagner-Spital Baumgartner Hohe, Vienna
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Odense University Hospital, Odense C, Denmark
- France (7):
  - Hopital Albert Michallon, Grenoble, Auvergne-Rhône-Alpes
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre de Lutte Contre le Cancer Francois Baclesse, Caen, Basse-normandie
  - Hopital Charles Nicolle, Rouen, Haute-normandie
  - Centre Hospitalier Universitaire Hopital Nord, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Intercommunal de Creteil, Créteil, Île-de-France Region
  - Hopital Tenon, Paris, Île-de-France Region
- Germany (6):
  - Universitatsklinik Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Kliniken der Stadt Koeln gGmbH - Krankenhaus Merheim, Cologne, North Rhine-Westphalia
  - Evangelische Lungenklinik Berlin, Berlin
  - Studiengesellschaft Haemato-Onkologie Hamburg Prof. Laack und Partner, Hamburg
- Hong Kong (3):
  - Tuen Mun Hospital, Tuenmen, New Territories
  - Queen Mary Hospital, Hong Kong
  - Queen Elizabeth Hospital, Kowloon
- Italy (13):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-cesena
  - Azienda Ospedaliera San Gerardo di Monza, Monza, Monza E Brianza
  - Centro di Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Istituto Oncologico di Bari Giovanni Paolo II, Bari
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Istituto Scientifico Universitario San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Tumori Napoli Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carita, Novara
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia, Perugia
  - Azienda Unita Sanitaria Locale di Ravenna, Ravenna
  - Policlinico Universitario Campus Bio-Medico, Roma
- Centre Hospitalier de Luxembourg - Hopital Municipal, Luxembourg, Luxembourg
- Netherlands (4):
  - Amphia Ziekenhuis - Locatie Langendijk Breda, Breda, North Brabant
  - Antoni van Leeuwenhoekziekenhuis, Amsterdam, North Holland
  - Isala Klinieken, Zwolle, Overijssel
  - Universitair Medisch Centrum Groningen, Groningen
- Radiumhospitalet, Oslo, Norway
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - OncoCare Cancer Centre, Singapore
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul
- Spain (12):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Teresa Herrera - Materno Infantil, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario Carlos Haya Malaga Instituto de Neurociencias Clinicas, Málaga
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Karolinska Universitetssjukhuset, Stockholm, Sweden
- University Hospital Zurich, Zurich, Switzerland
- Taiwan (5):
  - National Cheng Kung University, Tainan, Taipei
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (6):
  - Leicester Royal Infirmary, Leicester, England
  - University College London, London, England
  - Guy's and Saint Thomas' NHS Foundation Trust, London, England
  - Royal Marsden NHS Trust, London, England
  - Maidstone Hospital, Maidstone, England
  - The Christie NHS Foundation Trust, Manchester, England

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ahn MJ, Delmonte A, Ghosh S, Hochmair M, Yang TY, Yang JC, Han JY, Hansen KH, Wu Y, Wan Y, Lin HM, Kretz J, Hupf B, Kurec AM, Churchill EN, Fram RJ, Cabasag CJ, Goriya V, Zhao Y, Campelo MRG. Real-world treatment patterns and subsequent treatment effectiveness following frontline brigatinib in the ALTA-1L trial. Future Oncol. 2025 Dec;21(30):3935-3945. doi: 10.1080/14796694.2025.2592527. Epub 2025 Dec 18. PMID 41410381
- [Derived] Al Tawil A, McGrath S, Ristl R, Mansmann U. Addressing treatment switching in the ALTA-1L trial with g-methods: exploring the impact of model specification. BMC Med Res Methodol. 2024 Dec 20;24(1):314. doi: 10.1186/s12874-024-02437-6. PMID 39707229
- [Derived] Camidge DR, Kim HR, Ahn MJ, Yang JCH, Han JY, Hochmair MJ, Lee KH, Delmonte A, Garcia Campelo MR, Kim DW, Griesinger F, Felip E, Califano R, Spira A, Gettinger SN, Tiseo M, Lin HM, Gupta N, Hanley MJ, Ni Q, Zhang P, Popat S. Brigatinib Versus Crizotinib in Advanced ALK Inhibitor-Naive ALK-Positive Non-Small Cell Lung Cancer: Second Interim Analysis of the Phase III ALTA-1L Trial. J Clin Oncol. 2020 Nov 1;38(31):3592-3603. doi: 10.1200/JCO.20.00505. Epub 2020 Aug 11. PMID 32780660
- [Derived] Camidge DR, Kim HR, Ahn MJ, Yang JC, Han JY, Lee JS, Hochmair MJ, Li JY, Chang GC, Lee KH, Gridelli C, Delmonte A, Garcia Campelo R, Kim DW, Bearz A, Griesinger F, Morabito A, Felip E, Califano R, Ghosh S, Spira A, Gettinger SN, Tiseo M, Gupta N, Haney J, Kerstein D, Popat S. Brigatinib versus Crizotinib in ALK-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2027-2039. doi: 10.1056/NEJMoa1810171. Epub 2018 Sep 25. PMID 30280657
- [Derived] Gainor JF, Shaw AT. J-ALEX: alectinib versus crizotinib in ALK-positive lung cancer. Lancet. 2017 Jul 1;390(10089):3-4. doi: 10.1016/S0140-6736(17)31074-7. Epub 2017 May 10. No abstract available. PMID 28501139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 92 investigative sites in Australia, Hong Kong, Singapore, South Korea, Taiwan, Austria, Denmark, France, Germany, Italy, Luxembourg, Netherlands, Norway, Spain, Sweden, Switzerland, United Kingdom, Canada, and the United States of America from 26 May 2016 to 29 January 2021.
Pre-assignment Details: Participants with anaplastic lymphoma kinase and non-small-cell lung cancer (ALK+ NSCLC) who had not previously received an ALK-targeted tyrosine kinase inhibitor (TKI) were enrolled in 1:1 ratio to receive brigatinib 90 mg for 7 days followed by 180 mg or crizotinib 250 mg. Participants from crizotinib arm who experienced progressive disease (PD) or received radiotherapy to the brain in Randomized Phase were crossed over to receive brigatinib 90 mg/180 mg in the Crossover Phase.
Groups:
- Randomized Phase: Brigatinib 90 mg QD/180 QD: Brigatinib 90 mg, tablets, orally, once daily (QD) for first 7 days followed by 180 mg, orally, QD, in each 28-day cycle until disease progression (PD), intolerable toxicity, consent withdrawal, or death (The median duration of exposure was 34.86 months).
- Randomized Phase: Crizotinib 250 mg BID: Crizotinib 250 mg, tablets, twice daily (BID) in each 28-day cycle until disease progression, intolerable toxicity, consent withdrawal, or death (The median duration of exposure was 9.26 months).
- Crossover Phase: Brigatinib 90 mg QD/180 mg QD: Participants who experienced PD as assessed by the blinded Independent Review Committee (BIRC) or received radiotherapy to the brain while on 'Crizotinib 250 mg BID' therapy in Randomized Phase were crossed over. Following 10-day washout period, crossover participants received brigatinib 90 mg, tablets, orally, QD for first 7 days followed by 180 mg, tablets, orally, QD in each 28-day cycle up to end of the study (The median duration of exposure was 17.25 months).
Period: Randomized Phase
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Started | 137 | 138 | 0
Safety Analysis Set | 136 | 137 | 0
Completed | 20 | 84 | 0
Not Completed | 117 | 54 | 0
Not completed — Died | 41 | 29 | 0
Not completed — Withdrawal by Subject | 16 | 6 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Site Terminated by Sponsor | 58 | 16 | 0
Not completed — Reason not Specified | 1 | 1 | 0
Not completed — Never Treated | 1 | 1 | 0
Period: Crossover Phase
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Started | 0 | 0 | 65
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 55
Not completed — Died | 0 | 0 | 22
Not completed — Withdrew Consent | 0 | 0 | 9
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Site Terminated by Sponsor | 0 | 0 | 23

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all participants randomized to each regimen regardless of whether they tested ALK+, or whether they received study drug or adhered to the assigned dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Total
Number analyzed (Participants) | 137 | 138 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (13.46) | 58.6 (11.42) | 58.2 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 81 | 150
  Male | 68 | 57 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 59 | 49 | 108
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 76 | 86 | 162
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic, Latino or Spanish | 6 | 10 | 16
  Not Hispanic, Latino or Spanish | 131 | 128 | 259
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 2 | 5 | 7
  Hong Kong | 10 | 6 | 16
  Singapore | 5 | 1 | 6
  Korea, Republic Of | 29 | 28 | 57
  Taiwan, Province Of China | 12 | 9 | 21
  Austria | 5 | 4 | 9
  Denmark | 2 | 1 | 3
  France | 7 | 4 | 11
  Germany | 6 | 11 | 17
  Italy | 19 | 19 | 38
  Luxembourg | 1 | 0 | 1
  Netherlands | 5 | 6 | 11
  Norway | 0 | 2 | 2
  Spain | 14 | 17 | 31
  Sweden | 0 | 1 | 1
  Switzerland | 0 | 1 | 1
  United Kingdom | 10 | 8 | 18
  Canada | 0 | 2 | 2
  United States | 10 | 13 | 23
Global Health Status/Quality of Life (QoL) [Mean (Full Range); unit: score on a scale] — HRQoL:perceived quality of participant's life,includes self-reported multidimensional measures of physical,mental health.EORTC-QLQ-C30 contains 30 items across 5 functional scales(physical,role,cognitive,emotional,social),9 symptom scales(fatigue,nausea and vomiting,pain,dyspnea,sleep disturbance,appetite loss,constipation,diarrhea,financial difficulties),a global health status/QOL scale on 4 response levels(not at all,a little,quite a bit,very much),with 2 questions relying on a 7-point numeric rating scale.Raw scores converted into overall score of 0-100,lower scores indicate better QOL. Population: Number analyzed is number of participants with data available for global health status/QoL at Baseline.
  score on a scale
    number analyzed (Participants) | 131 | 131 | 262
    (all) | 60.432 [0.00 to 100.00] | 59.160 [0.00 to 100.00] | 59.796 [0.00 to 100.00]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS as assessed by Blinded Independent Review Committee (BIRC), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, was defined as the time interval from the date of randomization until the date of the first documented PD event. The data was censored for participants without a PFS event.
Time Frame: Up to end of study (Up to 56 months)
Population: ITT Population included all participants randomized to each regimen regardless of whether they tested ALK+, or whether they received study drug or adhered to the assigned dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 137 | 138 | 65
months | 24.016 [18.46 to 43.20] | 11.072 [9.13 to 13.01] | 16.821 [10.12 to 23.85]
Statistical Analysis 1: Comparison: Randomized Phase: Brigatinib 90 mg QD/180 QD vs Randomized Phase: Crizotinib 250 mg BID; Test type: Superiority; p < 0.0001, Log Rank — P-values are from a log-rank test stratified by randomization stratification factors (current; presence of intracranial central nervous system (iCNS) metastases at baseline and prior chemotherapy for locally advanced or metastatic disease); Hazard Ratio (HR) = 0.481, 95% CI 2-sided [0.35 to 0.66] — The hazard ratio was obtained using a Cox proportional hazards model with randomization stratification factors (current) as covariates

2. Secondary Outcome: Confirmed Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants who achieved Complete response (CR) or Partial responses (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) version (v). 1.1 criteria. CR is defined as disappearance of all extranodal target and non-target lesions. All pathological lymph nodes must have decreased to less than (<) 10 mm in short axis for target lesions and all lymph nodes must be non-pathological in size (<10 mm short axis), normalization of tumor marker level for non-target lesions. PR is at least a 30% decrease in SLD of target lesions, taking as reference baseline sum diameters.
Time Frame: Baseline up to end of treatment (Up to 36 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 137 | 138 | 65
percentage of participants | 74.5 [66.30 to 81.52] | 62.3 [53.68 to 70.42] | 56.9 [44.04 to 69.15]
Statistical Analysis 1: Comparison: Randomized Phase: Brigatinib 90 mg QD/180 QD vs Randomized Phase: Crizotinib 250 mg BID; Test type: Superiority; p = 0.0330, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.04 to 2.91] — Odds ratios and p-values were from a Cochran-Mantel-Haenszel test stratified by presence of intracranial central nervous system (iCNS) metastases at Baseline, and prior chemotherapy for locally advanced or metastatic disease (current strata)

3. Secondary Outcome: Confirmed Intracranial ORR (iORR)
Description: ORR was defined as percentage of participants who achieved CR or PR in the central nervous system (CNS) in randomized participants with intracranial CNS metastasis at baseline. CR is defined as disappearance of all extranodal target and non-target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis for target lesions and all lymph nodes must be non-pathological in size (<10 mm short axis), normalization of tumor marker level for non-target lesions. PR is at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to end of treatment (Up to 36 months)
Population: ITT Population included all participants randomized to each regimen regardless of whether they tested ALK+, or whether they received study drug or adhered to the assigned dose. Overall number of participants analyzed are the participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 47 | 49 | 42
percentage of participants | 66.0 [50.69 to 79.14] | 14.3 [5.94 to 27.24] | 35.7 [21.55 to 51.97]
Statistical Analysis 1: Comparison: Randomized Phase: Brigatinib 90 mg QD/180 QD vs Randomized Phase: Crizotinib 250 mg BID; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 13.56, 95% CI 2-sided [4.70 to 39.11] — Odds ratios and p-values were from a Cochran-Mantel-Haenszel test stratified by presence of prior chemotherapy for Locally advanced or metastatic disease at study entry (current strata)

4. Secondary Outcome: Intracranial Progression Free Survival
Description: Intracranial PFS as assessed by BIRC, is defined as the time from randomization until first CNS PD is documented, or death due to any cause. PD is SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest), the SLD must also demonstrate an absolute increase of at least 5 mm, and unequivocal progression of existing non-target lesions.
Time Frame: Baseline up to end of study (Up to 56 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 47 | 49 | 42
months | 23.951 [12.91 to 30.78] | 5.520 [3.71 to 7.52] | 24.542 [12.58 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Randomized Phase: Brigatinib 90 mg QD/180 QD vs Randomized Phase: Crizotinib 250 mg BID; Test type: Superiority; p < 0.0001, Log Rank — P-values are from a log-rank test stratified by randomization stratification factors (current; presence of iCNS metastases at baseline and prior chemotherapy for locally advanced or metastatic disease); Hazard Ratio (HR) = 0.293, 95% CI 2-sided [0.17 to 0.51] — The hazard ratio was obtained using a Cox proportional hazards model with prior chemotherapy for locally advanced or metastatic disease (current strata) as covariate

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: Baseline up to end of study (Up to 56 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 137 | 138 | 65
months | NA [NA to NA] — Median and 95% CI was not estimable due to fewer number of participants with events. | NA [NA to NA] — Median and 95% CI was not estimable due to fewer number of participants with events. | 35.023 [30.42 to NA] — Upper limit of 95% CI was not estimable due to fewer number of participants with events.

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response as assessed by BIRC, is defined as the time interval from the date that the criteria are first met for CR/PR (whichever is first recorded) until the first date that progressive disease (PD) is objectively documented. CR is defined as disappearance of all extranodal target and non-target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis for target lesions and all lymph nodes must be non-pathological in size (<10 mm short axis), normalization of tumor marker level for non-target lesions. PR is at least a 30 % decrease in the SLD of target lesions, taking as reference the baseline sum diameters. PD is SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest), the SLD must also demonstrate an absolute increase of at least 5 mm, and for non-target lesions, unequivocal progression of existing non-target lesions.
Time Frame: Baseline up to end of study (Up to 56 months)
Population: ITT Population included all participants randomized to each regimen regardless of whether they tested ALK+, or whether they received study drug or adhered to the assigned dose. Only responders were reported for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 102 | 86 | 37
months | 33.150 [1.84 to 50.60] | 13.832 [1.45 to 49.81] | 19.154 [1.97 to 33.15]

7. Secondary Outcome: Time to Response (TTR)
Description: Time to response as assessed by BIRC, assessment and is defined as the time interval from the date of randomization until the initial observation of CR or PR. CR is defined as disappearance of all extranodal target and non-target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis for target lesions and all lymph nodes must be non-pathological in size (<10 mm short axis), normalization of tumor marker level for non-target lesions. PR is at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to end of treatment (Up to 36 months)
Population: as for outcome 6
Measure: Median (Full Range); unit: months
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 137 | 138 | 65
months | 1.840 [1.02 to 29.47] | 1.873 [0.79 to 7.43] | 1.873 [0.20 to 18.33]

8. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control as assessed by BIRC, defined as percentage of randomized participants who have achieved CR, PR, or stable disease (SD) after randomization. CR defined as disappearance of all extranodal target and non-target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis for target lesions and all lymph nodes must be non-pathological in size (<10 mm short axis), normalization of tumor marker level for non-target lesions. PR: at least a 30% decrease in SLD of target lesions, taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD: SLD increased by at least 20% from the smallest value on study, SLD must also demonstrate an absolute increase of at least 5 mm, and unequivocal progression of existing non-target lesions.
Time Frame: Baseline up to end of treatment (Up to 36 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 137 | 138 | 65
percentage of participants | 85.4 [78.36 to 90.85] | 86.2 [79.34 to 91.50] | 73.8 [61.46 to 83.97]
Statistical Analysis 1: Comparison: Randomized Phase: Brigatinib 90 mg QD/180 QD vs Randomized Phase: Crizotinib 250 mg BID; Test type: Superiority; p = 0.8220, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.47 to 1.82] — Odds ratios and p-values were from a Cochran-Mantel-Haenszel test stratified by presence of iCNS metastases at Baseline, and prior chemotherapy for locally advanced or metastatic disease (current strata)

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product whether or not considered related to the medicinal product. Any worsening of a preexisting condition which is temporally associated with the use of the study drug (i.e., occurs after the first dose of study drug) is also an AE. TEAEs are defined as AEs starting/worsening on or after the first dose of study treatment and no later than the earliest of 30 days after the last dose of the treatment to which the participant was assigned, or the day before start of brigatinib therapy in crossover participant.
Time Frame: From first dose up to 30 days after last dose of study drug (Up to approximately 37 months)
Population: Treated Population included all participant who received at least 1 dose of study drug and served as basis of safety analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
Number analyzed (Participants) | 136 | 137 | 65
percentage of participants | 100 | 100 | 98.5

10. Secondary Outcome: Change From Baseline in Global Health Status/Quality of Life as Assessed by EORTC QLQ-C30 (Version 3.0)
Description: HRQoL: perceived quality of participant's life, includes self-reported multidimensional measures of physical and mental health. Patient-reported symptoms (PROs) and HRQoL will be collected by administering the european organisation for research and treatment of cancer (EORTC) quality of life (QLQ)-C30 questionnaire. EORTC-QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/QOL scale. The 30 items have 4 response levels (not at all, a little, quite a bit, and very much), with 2 questions relying on a 7-point numeric rating scale. Raw scores are converted into overall score ranging from 0 to 100, where lower scores indicate better QOL. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID
Number analyzed (Participants) | 104 | 53
score on a scale | 4.007 (25.7563) | -4.088 (27.4748)
Statistical Analysis 1: Comparison: Randomized Phase: Brigatinib 90 mg QD/180 QD vs Randomized Phase: Crizotinib 250 mg BID; Test type: Superiority; p = 0.0295, Mixed Models Analysis — p-values were obtained using mixed effects models stratified by presence of iCNS metastases at study entry, prior chemotherapy at Baseline; A mixed effect model is used with an unstructured covariance matrix; Least Square Mean Difference = 5.79, 95% CI 2-sided [0.58 to 11.00]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality - Up to 56 months; Serious and other adverse events - From first dose up to 30 days after last dose of study drug (Up to approximately 37 months)
Description: All Cause-mortality: ITT Population included all participants randomized to each regimen regardless of whether they tested ALK+, or whether they received study drug or adhered to the assigned dose. Serious and other (Non-serious): Treated Population included all participants who received ≥1 dose of study drug and served as basis of safety analysis. Crossover Population included participants from 'Crizotinib 250 mg BID' who crossed over to brigatinib following BIRC-assessed PD.
Arm/Group | Randomized Phase: Brigatinib 90 mg QD/180 QD | Randomized Phase: Crizotinib 250 mg BID | Crossover Phase: Brigatinib 90 mg QD/180 mg QD
All-Cause Mortality (participants affected / at risk) | 41/137 | 29/138 | 22/65
Serious Adverse Events (participants affected / at risk) | 56/136 | 53/137 | 24/65
Other Adverse Events (participants affected / at risk) | 132/136 | 135/137 | 63/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: Brigatinib 90 mg QD/180 QD (N=136) | Randomized Phase: Crizotinib 250 mg BID (N=137) | Crossover Phase: Brigatinib 90 mg QD/180 mg QD (N=65)
Pneumonia (Infections and infestations) | 6 | 5 | 4
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 3 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Cytomegalovirus Oesophagitis (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Listeriosis (Infections and infestations) | 0 | 1 | 0
Pleural Infection (Infections and infestations) | 0 | 1 | 1
Septic Shock (Infections and infestations) | 0 | 1 | 0
Sinusitis Fungal (Infections and infestations) | 0 | 1 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 3
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hodgkins Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1
Seizure (Nervous system disorders) | 1 | 1 | 2
Balance Disorder (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Memory Impairment (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Partial Seizures (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0
Vocal Cord Paralysis (Nervous system disorders) | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 2 | 0
Central Nervous System Lesion (Nervous system disorders) | 0 | 1 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 2 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0
Neutropenic Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis Ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 1 | 0 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 0 | 1
Asthenia (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1
Mucosal Inflammation (General disorders) | 1 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 0
Sudden Death (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 3 | 0
General Physical Health Deterioration (General disorders) | 0 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 1 | 0 | 0
Lipase Increased (Investigations) | 1 | 0 | 0
Transaminases Abnormal (Investigations) | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain Herniation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Performance Status Decreased (General disorders) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 2
Salmonella Sepsis (Infections and infestations) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intraventricular Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: Brigatinib 90 mg QD/180 QD (N=136) | Randomized Phase: Crizotinib 250 mg BID (N=137) | Crossover Phase: Brigatinib 90 mg QD/180 mg QD (N=65)
Upper Respiratory Tract Infection (Infections and infestations) | 18 | 12 | 6
Nasopharyngitis (Infections and infestations) | 12 | 15 | 5
Urinary Tract Infection (Infections and infestations) | 10 | 11 | 5
Pneumonia (Infections and infestations) | 10 | 5 | 6
Respiratory Tract Infection (Infections and infestations) | 7 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 12 | 8 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 16 | 28 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 6 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 11 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 11 | 0
Insomnia (Psychiatric disorders) | 14 | 12 | 7
Depression (Psychiatric disorders) | 5 | 8 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 4
Headache (Nervous system disorders) | 31 | 25 | 16
Dizziness (Nervous system disorders) | 23 | 29 | 12
Paraesthesia (Nervous system disorders) | 12 | 9 | 5
Dysgeusia (Nervous system disorders) | 5 | 20 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 9 | 0
Taste Disorder (Nervous system disorders) | 3 | 8 | 0
Vision Blurred (Eye disorders) | 7 | 14 | 0
Photopsia (Eye disorders) | 1 | 29 | 0
Visual Impairment (Eye disorders) | 1 | 23 | 0
Bradycardia (Cardiac disorders) | 10 | 22 | 0
Sinus Bradycardia (Cardiac disorders) | 7 | 11 | 0
Hypertension (Vascular disorders) | 44 | 12 | 15
Hypotension (Vascular disorders) | 3 | 10 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 9 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 49 | 29 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 26 | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 13 | 7 | 8
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 10 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 78 | 77 | 17
Nausea (Gastrointestinal disorders) | 44 | 81 | 11
Vomiting (Gastrointestinal disorders) | 30 | 59 | 9
Constipation (Gastrointestinal disorders) | 26 | 57 | 10
Abdominal Pain (Gastrointestinal disorders) | 18 | 20 | 0
Dyspepsia (Gastrointestinal disorders) | 15 | 23 | 0
Stomatitis (Gastrointestinal disorders) | 12 | 9 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 11 | 26 | 0
Dry Mouth (Gastrointestinal disorders) | 8 | 6 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 12 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 16 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 8 | 6
Rash (Skin and subcutaneous tissue disorders) | 25 | 4 | 6
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 13 | 3 | 5
Rash Erythematous (Skin and subcutaneous tissue disorders) | 9 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 8 | 6 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 8 | 5 | 9
Eczema (Skin and subcutaneous tissue disorders) | 8 | 3 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 35 | 22 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 17 | 9
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 20 | 15 | 17
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 15 | 11 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 11 | 11
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 12 | 10 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9 | 19 | 9
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Fatigue (General disorders) | 28 | 31 | 9
Pyrexia (General disorders) | 20 | 22 | 9
Asthenia (General disorders) | 18 | 26 | 8
Oedema Peripheral (General disorders) | 13 | 63 | 6
Non-Cardiac Chest Pain (General disorders) | 11 | 10 | 0
Malaise (General disorders) | 7 | 3 | 0
Influenza Like Illness (General disorders) | 6 | 11 | 10
Peripheral Swelling (General disorders) | 5 | 8 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 68 | 23 | 31
Aspartate Aminotransferase Increased (Investigations) | 35 | 36 | 17
Alanine Aminotransferase Increased (Investigations) | 31 | 49 | 11
Lipase Increased (Investigations) | 31 | 23 | 18
Amylase Increased (Investigations) | 25 | 13 | 14
Blood Alkaline Phosphatase Increased (Investigations) | 17 | 18 | 4
Blood Cholesterol Increased (Investigations) | 13 | 1 | 5
Blood Creatinine Increased (Investigations) | 8 | 20 | 0
Electrocardiogram Qt Prolonged (Investigations) | 8 | 8 | 5
Blood Lactate Dehydrogenase Increased (Investigations) | 7 | 5 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 5 | 8 | 0
Neutrophil Count Decreased (Investigations) | 3 | 14 | 0
Amylase Increased (Investigations) | 0 | 0 | 14
Blood Insulin Increased (Investigations) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT02737501/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT02737501/SAP_001.pdf